CLINICAL TRIAL: NCT06209060
Title: The Effect of Hammock Position and Nesting on the Comfort Level and Physiological Parameters of Preterm Babies
Brief Title: Hammock Position and Nesting in the Neonatal Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/85-58
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Behavior, Nesting; Behavior, Child
Keywords: position; comfort; behavior; hammock position; nesting; preterm
MeSH Terms: conditions — Nesting Behavior; Child Behavior; Behavior; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hammock Position Group (Experimental): Babies in the hammock position group will be placed in a hammock created by the researchers inside the incubator.
  Interventions: Behavioral: Hammock Position
- Nesting Group (Experimental): Babies in the nesting group will be placed in a nest created by the researchers within the incubator.
  Interventions: Behavioral: Nesting

INTERVENTIONS:
Behavioral: Hammock Position — Researchers will make a hammock by using a soft rectangular cotton cloth with ropes that pass through the circular openings of the incubator and are tied on the upper part of it. Babies will be placed in this hammock in a supine position with their extremities in the midline. The spine of the preterm neonate will support while arms and knees are flexed. Additionally, a small rectangular roller will be placed between the cervical and scapular region of the newborn in the hammock position to ensure that no hyperflexion or hyperextension position of the head occurs, which may impair respiratory function.
  Arms: Hammock Position Group
Behavioral: Nesting — In the nesting group, a nest will be made using rolls prepared with materials such as towels and blankets, and the baby will be placed in this nest. The baby's head and body will be positioned on the same axis, its extremities will be positioned in the midline, and its hands will be positioned close to its face.
  Arms: Nesting Group

SUMMARY:
This research aims to determine the effect of hammock position and nesting practices on the comfort level and physiological parameters of preterm babies.

DETAILED DESCRIPTION:
The study will be conducted with the randomized controlled experimental method. The sample size determined in the sample width analysis was determined as 72 babies (hammock position group: 36 babies; nesting group: 36 babies) with an effect size of 0.6, alpha error probability of 0.05, and a power value of 0.80. A sample of 72 preterm neonates will be randomly assigned into two equal groups. Neonates in the hammock position group will be placed in a hammock created by the researchers inside the incubator. Neonates in the nesting group will be placed in a nest created by the researchers within the incubator. Babies will be fed and their diapers changed before being positioned. These positions will be applied to babies for one hour every day for 5 consecutive days. Before positioning, the pulse oximeter device will be attached to the baby's foot, and its physiological parameters will be evaluated by remaining on the baby's foot for the duration of the positioning. During the one-hour position, no invasive procedures or diaper changes will be performed on the babies, the baby will not be touched, only observation will be made. The babies' comfort levels will be evaluated with the 'Newborn Comfort Behavior Scale' 5 minutes before positioning, at the 2nd, 20th, 40th, 60th minutes of positioning and 5 minutes after positioning, and their physiological parameters will be measured. The babies' comfort level will be evaluated independently by two observers.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies between 32-37 weeks of gestation
* The weight of the baby is 1500 grams and above,
* Postnatal age is 3 days or more,
* Preterm babies who have been in the Neonatal Intensive Care Unit for more than 24 hours,
* The baby is fed intermittently for more than 60 minutes,
* 30 minutes have passed since feeding,
* Do not perform procedures such as peripheral vascular access, blood collection, or gastric tube placement on the baby within the last hour before being taken into the study,
* Not applying phototherapy to the baby,
* No problems with the central nervous system such as cranial bleeding, convulsion, hypertonia,
* The baby does not have any congenital anomalies or respiratory distress,
* The baby does not receive oxygen support and is not connected to a respirator.

Exclusion Criteria:

* Babies younger than 32 weeks of gestation and older than 37 weeks of gestation
* The baby's weight is below 1500 grams,
* Postnatal age is less than 3 days,
* Preterm babies who have been in the Neonatal Intensive Care Unit for less than 24 hours,
* The baby is fed at intervals of less than 60 minutes,
* Less than 30 minutes have passed since feeding,
* Performing procedures such as peripheral vascular access, blood collection, and gastric tube placement on the baby within the last hour before being taken into the study,
* Applying phototherapy to the baby,
* Having a problem with the central nervous system such as cranial hemorrhage, convulsion, hypertonia,
* Presence of the baby's congenital anomaly or respiratory distress,
* The baby receives oxygen support and is connected to a respirator.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Comfort Level | 5 minutes before positioning the neonate, at the 2nd, 20th, 40th, 60th minute of positioning the neonate, 5 minutes after positioning the neonate.
  The preterm babies' comfort levels will be determined using the Newborn Comfort Behavior Scale (COMFORTneo). COMFORTneo is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. In addition to determining comfort, the Newborn Comfort Behavior Scale allows nurses to evaluate the baby's pain and distress. It has been stated that the lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6 and the highest score is 30. COMFORTneo score values under 13 indicate no pain or stress, values between 14 and 21 indicate moderate pain or stress, and values between 22 and 30 indicate severe pain or stress.

SECONDARY OUTCOMES:
Heart Rate | 5 minutes before positioning the neonate, at the 2nd, 20th, 40th, 60th minute of positioning the neonate, 5 minutes after positioning the neonate.
  The researchers recorded the neonates' heart rate from the ECG monitor
Respiration Rate | 5 minutes before positioning the neonate, at the 2nd, 20th, 40th, 60th minute of positioning the neonate, 5 minutes after positioning the neonate.
  The researchers recorded the neonates' respiration rate from the ECG monitor
Oxygen Saturation | 5 minutes before positioning the neonate, at the 2nd, 20th, 40th, 60th minute of positioning the neonate, 5 minutes after positioning the neonate.
  The researchers recorded the neonates' oxygen saturation from the ECG monitor

CONTACTS AND LOCATIONS:
Overall Officials: Selmin Köse, PhD, Principal Investigator — Biruni University
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No